CLINICAL TRIAL: NCT05573815
Title: An Open Label, Single-Center and Random-Selection Retrospective Pivotal Study of Clinical Decision Support System for Brain Metastasis Using Brain MR Images
Brief Title: Evaluation of Clinical Decision Support System for Brain Metastasis Using Brain MR Images
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heuron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HR-BM-01
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive group (Experimental): A patient diagnosed with brain metastasis after a brain MR
  Interventions: Device: BT-M01
- Negative group (Experimental): A normal person or a patient not diagnosed with brain metastasis after a brain MR
  Interventions: Device: BT-M01

INTERVENTIONS:
Device: BT-M01 — Clinical decision support system for detecting brain metastasis

SUMMARY:
BT-M01 is a software that has been pre-learned based on a brain metastasis detection model using brain MR images, and clinical decision support system for brain metastasis by automatically analyzing brain MR images by assisting the medical team.

The specific aims of this study are to evaluate efficacy of BT-M01 for brain metastasis compared to the sensitivity and false positive rates of radiologists group.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years old
* Brain MR acquired
* Positive group: A patient diagnosed with brain metastasis after a brain MR
* Negative group: A normal person or a patient not diagnosed with brain metastasis after a brain MR

Exclusion Criteria:

* Poor or incomplete brain MR image quality
* A patient with other pathological lesion in brain
* A patients with a history of primary brain tumors

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and false positive rates of BT-M01 | Within 4 weeks after enrollment
  Sensitivity and false positive rates of BT-M01 in detection of brain metastasis based on golden standards

SECONDARY OUTCOMES:
Positive predictive values of BT-M01 | Within 4 weeks after enrollment
  Positive predictive values of BT-M01 in detection of brain metastasis based on golden standards
Sensitivity and Positive predictive values of BT-M01 by primary cancer | Within 4 weeks after enrollment
  Sensitivity and positive predictive values of BT-M01 in detection of brain metastasis based on golden standards by primary cancer
Dice coefficient of BT-M01 | Within 4 weeks after enrollment
  Dice coefficient of BT-M01 in detection of brain metastasis based on golden standards

CONTACTS AND LOCATIONS:
Overall Officials: Ji Eun Park, M.D.pH.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Song-pa Gu, South Korea

IPD SHARING:
Plan to Share IPD: No